CLINICAL TRIAL: NCT07230769
Title: Impact of Bougie Diameter on Outcomes in Laparoscopic Sleeve Gastrectomy - A Randomized Controlled Trial
Brief Title: Bougie Diameter on Outcomes in Laparoscopic Sleeve Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Mohamed Hany Ashour, Professor of General surgery, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Bougie Diameter Outcomes LSG
Record Dates: First submitted 2025-09-21; First posted 2025-11-17 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Bariatric Sleeve Gastrectomy
Keywords: Bougie Diameter; Outcomes in Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: This is a prospective, randomized, double-blind controlled trial (RCT) comparing two different bougie diameters in laparoscopic sleeve gastrectomy. The study will involve:
  * Group1 : LSG performed using a >40-Fr diameter calibration bougie
  * Group2 : Standard care using 36-Fr diameter calibration bougie
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 : LSG performed using a >40-Fr diameter calibration bougie (Active Comparator): LSG performed using a >40-Fr diameter calibration bougie
  Interventions: Device: Bougie (>40-Fr)
- Group2 : Standard care using 36-Fr diameter calibration bougie (Active Comparator): Standard care using 36-Fr diameter calibration bougie
  Interventions: Device: Bougie (36-Fr)

INTERVENTIONS:
Device: Bougie (>40-Fr) — * Product: MID-TUBE orogastric calibration tube (Médical Innovation Development S.A.S, ref. MID131)
  * Classification: CE-marked class IIa medical single-use device
  * Length: 70 cm
  * Material: Medical silicon rubber, latex-free
  Arms: Group1 : LSG performed using a >40-Fr diameter calibration bougie
Device: Bougie (36-Fr) — * Various manufacturers' single-use devices
  * All devices CE-marked and used per manufacturer instructions
  * Specific size selection based on center standard care protocols
  Arms: Group2 : Standard care using 36-Fr diameter calibration bougie

SUMMARY:
Laparoscopic sleeve gastrectomy (LSG) has become an increasingly popular bariatric procedure since its first performance by Hess and Hess in 1988 as a component of the biliopancreatic diversion-duodenal switch (BPD-DS) procedure, which was modified from Scopinaro's biliopancreatic diversion (BPD) and DeMeester's technique. In the early part of the twenty-first century, it was popularized as a first-step intervention before BPD or gastric bypass in the super obese and high-risk group of patients by Regan et al. Due to the unexpected good results in terms of weight loss and resolution of comorbidities, coupled with the simplicity of performing the procedure requiring intervention on only the stomach, sleeve gastrectomy gained status as a stand-alone bariatric procedure as demonstrated by Baltasar et al.

The basic principle of LSG is to create a narrow stomach along the lesser curvature, depending on the left gastric artery, using a calibration bougie as a template to perform a vertical partial gastrectomy, resecting the greater curvature and fundus of the stomach according to the International Sleeve Gastrectomy Expert Panel Consensus Statement by Rosenthal et al. The procedure has demonstrated excellent outcomes in terms of weight loss and comorbidity resolution, making it one of the most commonly performed bariatric procedures worldwide according to the IFSO Worldwide Survey by Angrisani et al.

Bougie Size Considerations and Rationale The selection of an appropriate bougie size during laparoscopic sleeve gastrectomy represents a critical technical decision that significantly influences both immediate surgical outcomes and long-term patient results. Calibration bougies serve as internal templates to standardize the gastric sleeve diameter and ensure consistent sleeve geometry across different surgeons and institutions, as described by Parikh et al.

The diameter of the bougie directly determines the final gastric volume and the degree of restriction achieved, which in turn affects weight loss efficacy, food tolerance, and complication rates.

Bougie sizes in current clinical practice typically range from 32-French (Fr) to 50-Fr, with most centers utilizing sizes between 34-Fr and 42-Fr according to the survey by Gagner et al. Small bougie sizes (32-36-Fr) create a more restrictive sleeve with potentially enhanced weight loss but may be associated with increased risks of stenosis, food intolerance, and gastroesophageal reflux disease as reported by Sakran et al.

Medium bougie sizes (38-42-Fr) represent a compromise between restriction and safety, offering adequate weight loss while maintaining acceptable complication rates as demonstrated by Weiner et al. Large bougie sizes (44-50-Fr) provide greater sleeve capacity with improved food tolerance and potentially reduced leak rates, though concerns exist regarding long-term weight loss maintenance according to Abdallah et al.

The rationale for comparing different bougie sizes stems from the ongoing debate regarding the optimal balance between surgical efficacy and safety. Recent meta-analyses have suggested that larger bougie sizes may be associated with reduced gastric leak rates without significantly compromising weight loss outcomes. However, the majority of existing evidence comes from retrospective observational studies with inherent limitations including selection bias, confounding variables, and lack of standardized outcome measures as noted by Shi et al. The current study aims to provide definitive prospective evidence comparing small (36-Fr) versus X large (larger than 40-Fr) bougie sizes in a randomized controlled trial design.

Furthermore, the impact of bougie size on comorbidity resolution remains inadequately studied. Bariatric surgery has demonstrated remarkable efficacy in resolving obesity-related comorbidities, with diabetes remission rates ranging from 53% to 63% as reported by Schauer et al. and hypertension resolution rates varying from 8% to 50% depending on the specific criteria used according to Sjöström et al. The relationship between sleeve geometry, as determined by bougie size, and comorbidity resolution mechanisms requires further investigation to optimize patient outcomes and surgical technique selection.

DETAILED DESCRIPTION:
Hypothesis

The investigators hypothesize that the use of a larger calibration bougie (> 40-Fr) during laparoscopic sleeve gastrectomy will significantly reduce the incidence of postoperative gastric leak compared to standard smaller bougie sizes (36-Fr), without compromising weight loss outcomes or quality of life measures.

Hypotheses Tools

1. Quality of Life Hypothesis: Patients undergoing LSG with > 40-Fr bougie will demonstrate equivalent or superior quality of life outcomes as measured by the Moorehead-Ardelt Quality of Life Questionnaire II (MA-II) compared to those with smaller bougie sizes at 1-month, 6-months and 1-year follow-up.
2. Nutritional Tolerance Hypothesis: Larger bougie diameter (> 40-Fr) will result in improved food tolerance as assessed by the Suter et al. food tolerance questionnaire, leading to better nutritional outcomes and reduced gastrointestinal symptoms.
3. Weight Loss Hypothesis: Despite the larger gastric remnant created by the > 40-Fr bougie, total weight loss percentage (%TWL) at 6 months and 1 year will be non-inferior to that achieved with smaller bougie sizes, with the primary endpoint being ≥20% TWL at 1 year.
4. Complication Hypothesis: The use of >40-Fr bougie will be associated with a lower overall complication rate as classified by the Clavien-Dindo classification system, particularly for grades III-V complications requiring surgical intervention or resulting in life-threatening consequences.
5. Recovery Hypothesis: Patients in the >40-Fr bougie group will experience reduced postoperative pain as measured by Visual Analog Scale (VAS) scores and shorter hospital length of stay compared to the control group.
6. Upper Gastrointestinal Hypothesis: Upper gastrointestinal evaluation at 1 year will demonstrate equivalent or improved anatomical and functional outcomes in the >40-Fr group, with reduced incidence of strictures, gastroesophageal reflux disease, and other upper GI complications.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged between 18 and 70 years undergoing LSG as a primary bariatric procedure
2. Body mass index (BMI) criteria according to 2022 ASMBS/IFSO guidelines:

   * BMI ≥35 kg/m² regardless of presence, absence, or severity of comorbidities, OR
   * BMI 30-34.9 kg/m² (Class I obesity) with metabolic disease and inadequate response to nonsurgical methods, including:

     * Type 2 diabetes mellitus
     * Arterial hypertension
     * Dyslipidemia
     * Obstructive sleep apnea syndrome and other severe respiratory disorders
     * Cardiovascular disease (coronary artery disease, heart failure, atrial fibrillation)
     * Asthma
     * Fatty liver disease and nonalcoholic steatohepatitis
     * Chronic kidney disease
     * Polycystic ovarian syndrome
     * Infertility
     * Pseudotumor cerebri
     * Bone and joint diseases
3. Decision for bariatric surgery approved after multidisciplinary team discussion
4. Written informed consent obtained
5. Ability to complete questionnaires and attend follow-up visits
6. Stable weight (±5% for 3 months before surgery)
7. Normal preoperative upper gastrointestinal endoscopy or findings limited to:

   * Los Angeles (LA) Classification Grade A reflux esophagitis (minimal mucosal breaks <5mm)
   * Mild gastritis without active ulceration
8. Negative or minimal gastroesophageal reflux symptoms (GERD-Q score ≤8)

Exclusion Criteria:

1. History of previous gastric surgeries or bariatric procedures
2. American Society of Anesthesiologists (ASA) score >4
3. Ongoing pregnancy or planned pregnancy within the study period
4. Significant esophageal and gastric pathology, including:

   * Los Angeles (LA) Classification Grade B, C, or D reflux esophagitis
   * Hiatal hernia or any paraesophageal hernia
   * Barrett's esophagus of any length
   * Active peptic ulcer disease
   * Gastric polyps >1cm or suspicious lesions
5. Severe gastroesophageal reflux disease is defined as:

   * GERD-Q score >8
   * Daily proton pump inhibitor (PPI) dependency with breakthrough symptoms
   * Endoscopic evidence of LA Grade B, C, or D esophagitis
6. Coagulation disorders or anticoagulation therapy that cannot be safely discontinued
7. Known silicon hypersensitivity or allergies to bougie materials
8. Active substance abuse or psychiatric conditions that may impair compliance

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Gastric Leak Diagnosis and Classification | within 3 months postoperatively
  The diagnosis of gastric leak must be fulfilled with any of the following criteria within 3 months postoperatively according to Benedix et al.:
  1. Morphologic examination with contrast studies:
     * Abdominal CT scan with oral contrast showing extravasation
     * Upper gastrointestinal swallow studies demonstrating contrast leak
     * Abnormal perigastric pneumoperitoneum on imaging
  2. Surgical evidence:
     * Direct visualization of staple-line disruption during exploratory re-intervention
     * Exit of methylene blue dye through drainage during postoperative course
     * Endoscopic visualization of staple-line defect
  3. Endoscopic evidence:
     * Extravasation of contrast during endoscopy with C-arm fluoroscopy
     * Direct endoscopic visualization of gastric perforation or staple-line dehiscence
  Leak Classification System:
  * Type I (Early): 0-7 days postoperatively
  * Type II (Intermediate): 8-30 days postoperatively
  * Type III (Late): >30 days postoperatively

SECONDARY OUTCOMES:
Quality of Life Assessment - Moorehead-Ardelt Quality of Life Questionnaire II (MA-II) | will be administered at baseline, 1 month, 6 months, and 1 year postoperatively
  This validated instrument specifically designed for bariatric surgery patients evaluates six domains of quality of life:
  1. Self-Esteem: Assessment of patient's self-perception and confidence levels
  2. Physical Activity: Evaluation of exercise capacity and physical function
  3. Social Contacts: Assessment of social interactions and relationships
  4. Work Performance: Evaluation of occupational capacity and productivity
  5. Sexual Interest: Assessment of sexual function and interest
  6. Eating Behavior: Evaluation of eating patterns and food-related behaviors
  Each domain is scored from -3 to +3 points, with total MA-II Score Range: -18 to +18 points.
  Score interpretation:
  * Very poor quality of life: -18 to -9 points
  * Poor quality of life: -8 to -3 points
  * Fair quality of life: -2 to +2 points
  * Good quality of life: +3 to +8 points
  * Very good quality of life: +9 to +18 points
Food Tolerance Assessment - Suter Questionnaire | will be administered at 1, 3, 6, and 12 months postoperatively.
  The questionnaire evaluates:
  1. Overall Satisfaction with Food Intake (0-3 points):
     * 0 = Cannot eat normal food
     * 1 = Eats small amounts of normal food
     * 2 = Eats normal food with some restrictions
     * 3 = Eats normal food without restrictions
  2. Food Tolerance Score (0-24 points): Assessment of tolerance to 8 food categories:
     * Meat
     * Salad/raw vegetables
     * Fresh fruits
     * Bread
     * Rice/pasta
     * Vegetables
     * Dairy products
     * Liquids
     Each food scored 0-3 points:
     * 0 = Cannot eat at all
     * 1 = Can eat small amounts with difficulty
     * 2 = Can eat moderate amounts with some difficulty
     * 3 = Can eat normal amounts without difficulty
  3. Eating Behavior Assessment:
     * Eating frequency per day
     * Time required for meals
     * Chewing adequacy
     * Presence of food aversion
  Total Suter Score Range: 0-27 points
  * Excellent tolerance: 24-27 points
  * Good tolerance: 21-23 points
  * Fair tolerance: 18-20 points
  * Poor tolerance: <18 points
Weight Loss Assessment - Total Weight Loss Percentage (%TWL) | Baseline (preoperative) then 1, 3, 6, 12 months postoperative.
  Calculation Formula: %TWL = [(Initial weight - Current weight) / Initial weight] × 100 (weight is measured in kilograms Kg)
  Success Criteria according to Eisenberg et al.:
  * Adequate weight loss: ≥20% TWL at 12 months
  * Good weight loss: ≥25% TWL at 12 months
  * Excellent weight loss: ≥30% TWL at 12 months
Postoperative Nausea and Vomiting Assessment | Time Points: - 2 hours postoperatively - 6 hours postoperatively - 24 hours postoperatively - 48 hours postoperatively - Day 3 postoperatively
  Assessment Tool: Modified Postoperative Nausea and Vomiting (PONV) Scale according to Apfel et al.
  Nausea Assessment (0-10 scale):
  * 0 = No nausea
  * 1-3 = Mild nausea
  * 4-6 = Moderate nausea
  * 7-10 = Severe nausea
  Vomiting Assessment:
  * Number of vomiting episodes per 24-hour period
  * Volume of vomitus (estimated) (Volume is measured in milliliters mL)
  * Character of vomitus (bilious, food particles, blood)
  Antiemetic Usage:
  * Antiemetic administered
  * Dosage and frequency
  * Time to administration
  * Effectiveness assessment
Pain Assessment - Visual Analog Scale (VAS) | Assessment Schedule: - Immediate postoperative: Every 2 hours for first 24 hours - Postoperative day 1-2: Every 6 hours - Day 3 postoperatively: Final assessment - Follow-up visits: 1 week, 1 month
  VAS Pain Scale: 100mm horizontal line with anchors according to Hawker et al.
  * 0mm = "No pain"
  * 100mm = "Worst possible pain"
  Pain Categories:
  * No pain: 0-4mm
  * Mild pain: 5-44mm
  * Moderate pain: 45-74mm
  * Severe pain: 75-100mm
  Additional Pain Assessments:
  * Location of pain (incisional, abdominal, shoulder)
  * Pain character (sharp, dull, cramping)
  * Pain interference with activities
  * Analgesic requirements and effectiveness
Hospital Length of Stay Assessment | Baseline till Day 3 postoperatively.
  Measurement Parameters:
  * Admission time: Date and time of hospital admission
  * Surgery time: Date and time of procedure completion
  * Discharge time: Date and time of hospital discharge
  * Total length of stay: Hours from admission to discharge
  * Postoperative length of stay: Hours from surgery completion to discharge
  * Need for re-admission
  Discharge Criteria:
  * Stable vital signs for 6 hours
  * Adequate pain control with oral medications
  * Tolerance of clear liquids without nausea/vomiting
  * Ambulation without assistance
  * No signs of complications
  * Patient understanding of discharge instructions
Postoperative Complications - Clavien-Dindo Classification | within 30 days
  All complications within 30 days will be classified using the Clavien-Dindo system Grade I: Any deviation from normal postoperative course without need for pharmacological, surgical, endoscopic, or radiological interventions
  Grade II: Requiring pharmacological treatment with drugs other than allowed for Grade I complications
  Grade III: Requiring surgical, endoscopic, or radiological intervention
  * Grade IIIa: Intervention not under general anesthesia
  * Grade IIIb: Intervention under general anesthesia
  Grade IV: Life-threatening complications requiring intensive care management
  * Grade IVa: Single organ dysfunction
  * Grade IVb: Multi-organ dysfunction
  Grade V: Death of patient
  Suffix "d": Added if patient suffers from complication at discharge (e.g., Grade IIId)
Comorbidity Resolution Assessment | Assessment Time Points: 6 months and 12 months postoperatively
  The evaluation of comorbidity resolution and improvement will be conducted according to the standardized outcomes reporting criteria established by the American Society for Metabolic and Bariatric Surgery (ASMBS) Clinical Issues Committee, as published by Brethauer et al. This standardized approach ensures consistency with current best practices and facilitates comparison with other bariatric surgery studies.
  Type 2 Diabetes Mellitus:
  * Complete remission: HbA1c <6.0% without antidiabetic medications for ≥1 year
  * Partial remission: HbA1c 6.0-6.4% without antidiabetic medications for ≥1 year
  * Improvement: Reduction in HbA1c ≥1% or reduction in antidiabetic medications
  * No change: <1% change in HbA1c and same medications
  * Worsening: Increase in HbA1c or need for additional medications
Comorbidity Resolution Assessment | Assessment Time Points: 6 months and 12 months postoperatively
  The evaluation of comorbidity resolution and improvement will be conducted according to the standardized outcomes reporting criteria established by the American Society for Metabolic and Bariatric Surgery (ASMBS) Clinical Issues Committee, as published by Brethauer et al. This standardized approach ensures consistency with current best practices and facilitates comparison with other bariatric surgery studies.
  Arterial Hypertension:
  * Resolution: Blood pressure <140/90 mmHg without antihypertensive medications
  * Improvement: Reduction in number or dosage of antihypertensive medications
  * No change: Same blood pressure control with same medications
  * Worsening: Need for additional medications or poor control
Comorbidity Resolution Assessment | Assessment Time Points: 6 months and 12 months postoperatively
  The evaluation of comorbidity resolution and improvement will be conducted according to the standardized outcomes reporting criteria established by the American Society for Metabolic and Bariatric Surgery (ASMBS) Clinical Issues Committee, as published by Brethauer et al. This standardized approach ensures consistency with current best practices and facilitates comparison with other bariatric surgery studies.
  Dyslipidemia:
  * Resolution: Normal lipid profile without lipid-lowering medications
  * Improvement: Improvement in lipid parameters or reduction in medications
  * No change: Stable lipid profile with same medications
  * Worsening: Deterioration in lipids or need for additional medications
Comorbidity Resolution Assessment | Assessment Time Points: 6 months and 12 months postoperatively
  The evaluation of comorbidity resolution and improvement will be conducted according to the standardized outcomes reporting criteria established by the American Society for Metabolic and Bariatric Surgery (ASMBS) Clinical Issues Committee, as published by Brethauer et al. This standardized approach ensures consistency with current best practices and facilitates comparison with other bariatric surgery studies.
  Obstructive Sleep Apnea:
  * Resolution: Normal sleep study without CPAP therapy
  * Improvement: Reduced AHI or decreased CPAP pressure requirements
  * No change: Stable sleep study parameters
  * Worsening: Increased AHI or higher CPAP pressure requirements
Upper Gastrointestinal Evaluation | Mandatory 1-Year Upper GI Assessment GERD-Q Questionnaire Administration Timeline: - Preoperative: (baseline) - 1 month postoperative - 3 months postoperative - 6 months postoperative - 12 months postoperative
  Mandatory 1-Year Upper GI Assessment:
  1. Upper Gastrointestinal Endoscopy:
     * Systematic evaluation of esophagus, gastroesophageal junction, and gastric sleeve
     * Los Angeles (LA) Classification reassessment for reflux esophagitis
  2. GERD Symptom Reassessment:
     * GERD-Q questionnaire readministration
     * Arabic GERD-Q questionnaire for Arabic-speaking patients
     * Comparison with preoperative GERD-Q scores
     * Documentation of PPI usage changes from baseline
     * Assessment of new or worsening reflux symptoms
     * Evaluation of extraesophageal symptoms
  3. Upper GI Outcome Classification:
     * Improved: Reduction in GERD-Q score ≥2 points from baseline and/or improvement in LA grade
     * Stable: GERD-Q score change <2 points and stable LA grade
     * Worsened: Increase in GERD-Q score ≥2 points and/or progression in LA grade
     * New-onset GERD: Development of GERD-Q score >8 in previously asymptomatic patients
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment
  - Complete blood count (CBC)
  Normal ranges for a Complete Blood Count (CBC) vary by age, sex, and even the laboratory performing the test, but generally, adult normal ranges include:
  * Red Blood Cell Count (RBC): ~4.2-6.1 million cells/mcL (in number of cells per microliter)
  * White Blood Cell Count (WBC): ~4,500-11,000 cells/mcL (in number of cells per microliter)
  * Hemoglobin: ~12-18 g/dL (in grams per deciliter)
  * Platelets: ~150,000-450,000/mcL (in number of cells per microliter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Comprehensive metabolic panel Normal ranges for a comprehensive metabolic panel (CMP) can vary by laboratory, but generally include values for glucose (70-100 mg/dL), calcium (8.5-10.2 mg/dL), blood urea nitrogen (BUN) (6-20 mg/dL), and creatinine (0.6-1.3 mg/dL). The CMP also includes liver function tests such as albumin (3.4-5.4 g/dL), total protein (6.0-8.3 g/dL), alkaline phosphatase (20-130 U/L), ALT (4-36 U/L), AST (8-33 U/L), and total bilirubin (0.1-1.2 mg/dL).
  (measured in Grams or milligrams per deciliter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Lipid profile Normal lipid profile levels in mg/dL for adults are generally Total Cholesterol below 200, LDL (bad) Cholesterol below 100, HDL (good) Cholesterol 40 or higher for men and 50 or higher for women, and Triglycerides below 150.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Hemoglobin A1c A normal HbA1c range is generally considered below 5.7%, which indicates healthy blood sugar levels. The ranges for prediabetes and diabetes are 5.7% to 6.4% and 6.5% or higher, respectively. These results reflect average blood sugar levels over the past 2-3 months and are used to monitor, screen, and diagnose diabetes and prediabetes.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Thyroid function tests (free T4) Normal thyroid function test values vary by lab, age, and pregnancy status, but a typical range for adults is 9.0-25.0 pmol/L for free T4. (measured in picomoles per liter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment: - Thyroid function tests (Serum TSH) Normal thyroid function test values vary by lab, age, and pregnancy status, but a typical range for adults is 0.4-4.0 mIU/L for TSH. (measured in milli international unit per liter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Vitamin B12 Normal values for serum vitamin B12 typically fall in the range of 180-914 pg/mL. (measured in picograms per milliliter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Serum Folate Normal values for serum folate is around 4.0 ng/mL. (measured in nanograms per milliliter)
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - 25-hydroxyvitamin D Normal values for a 25-hydroxyvitamin D test vary, but generally, sufficiency is considered to be 20-50 ng/mL (50-125 nmol/L). Levels below 20 ng/mL (50 nmol/L) may indicate insufficiency, while levels below 10 ng/mL (25 nmol/L) often signify deficiency.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Iron studies (ferritin, transferrin saturation, TIBC) Serum Iron: Measures the amount of iron in the blood. Males: 50-150 mcg/dL (8.95-26.85 micromol/L) Females: 35-145 mcg/dL (6.26-25.95 micromol/L) Total Iron-Binding Capacity (TIBC): Measures the blood's ability to attach to iron.
  General Range: 250-450 mcg/dL (45-81 micromol/L) Transferrin Saturation: The percentage of transferrin (a protein that carries iron) that is saturated with iron.
  Males: 20-50% Females: 15-45% Ferritin: Measures the body's iron stores. Men: 30-300 ng/mL Women: 20-200 ng/mL
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Albumin and prealbumin Normal adult albumin levels are typically 3.5 to 5.5 g/dL, while normal adult prealbumin levels are usually 15 to 36 mg/dL.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Parathyroid hormone (PTH) Normal parathyroid hormone (PTH) levels typically fall between 10 and 65 pg/mL.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Calcium and phosphorus Normal serum calcium levels for adults are roughly 8.6-10.3 mg/dL, while normal phosphorus levels are approximately 2.5-4.5 mg/dL.
Nutritional and Laboratory Assessment | within 1,6,12 months preoperatively.
  Baseline Assessment:
  - Magnesium and zinc levels Normal magnesium levels are typically 1.7 to 2.2 mg/dL. Normal zinc levels, however, are more variable, with studies showing ranges such as 71.26-108.53 µg/dL in one population and 60.82-96.13 µg/dL in another.

CONTACTS AND LOCATIONS:
Locations (1):
- The surgical department of Medical Research Institute Hospital, Alexandria University, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
FAIR data of this study can be requested. All will be saved in the Castor Electronic data capture system.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Whole study period
Access Criteria: Ask contact person (Email the Principal investigator).